CLINICAL TRIAL: NCT01974128
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Cardiovascular Effects of Autologous Adipose-Derived Stromal Cells Implantation by a Catheter Delivery System and/or Intravenously In Patients During the Acute Recovery Phase of ST-Elevation Myocardial Infarction
Brief Title: Study to Assess the Safety and Cardiovascular Effects of Autologous Adipose-Derived Stromal Cells Implantation In Patients During the Acute Recovery Phase of ST-Elevation Myocardial Infarction
Acronym: Acute MI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ME-AMI-001
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-03

CONDITIONS: Acute Myocardial Infarction
Keywords: MI
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ASC isolation and implantation — This trial will study ASC implantation using a catheter delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The injection catheter will be used for delivery of the ASCs therapy

SUMMARY:
The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe? and 2) Is treatment effective in improving cardiac function and clinical outcomes?

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate in patients recovering from acute myocardial infarction (< 8 days after the index infarction) both the safety profile of intramyocardial ASCs and the preliminary efficacy of ASCs therapy.

This will be an open-label, non-randomized patient sponsored multi-center study of ASC implantation using a catheter delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The injection catheter will be used for delivery of the ASCs therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Defined acute myocardial infarction <8 days from screening
* Left ventricular ejection fraction at screening of ≤ 50%, with 2 or more contiguous areas of severe wall motion abnormality on resting echocardiography.
* Patients must have a minimum myocardial wall thickness of 5mm
* Need or feasibility for re-vascularization has been ruled out by coronary angiogram or noninvasive stress testing.
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* NYHA CHF Class 4
* Severe valvular or other non-ischemic myocardial disease.
* Mechanical complications of the index acute myocardial infarction including but not limited to rupture of the mitral valve with resultant development of mitral regurgitation, rupture of the left ventricular free wall and rupture of the interventricular septum.
* Active infectious disease and/or known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis. If the panel includes antibodies to the HBV-cAg and HBV-sAg, then an expert will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection within one week of enrollment.
* Cerebrovascular accident within 6 months prior to study entry
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Improvement | 6 months
  Autologous ASCs therapy will be considered effective for post-myocardial infarction patients if there is an improvement in:
  * Absolute LVEF
  * Changes in LVEF from baseline to 6 months
  * MI size
  * Regional wall thickness and thickening in all segments
  * LV-end systolic volume (LV-ESV)
  * LV-end diastolic volume (LV-EDV)
  * Change in perfusion defect after revascularization to six months as measured by:
    * Echocardiography
    * Scintigraphy

SECONDARY OUTCOMES:
Primary Safety Objective | 6 months
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ageless Institute, Miami, Florida, United States